CLINICAL TRIAL: NCT02406547
Title: Randomised Tandem Colonoscopy of Narrow Band Imaging (NBI) and White Light Endoscopy in Patients With Serrated Lesions
Brief Title: Study of Narrow Band Imaging in the Characterization of Serrated Lesions
Acronym: CROMOSER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Fausto Riu, MD, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: CROMOSER
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Serrated Polyps; Sessile Serrated Adenoma; Colorectal Neoplasms
Keywords: Serrated lesion; sessile serrated adenoma; Narrow Band Imaging; Colonoscopy; colorectal neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Narrow Band Imaging

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- WLE-NBI (Experimental): Participants will be evaluated by same endoscopist, back-to-back tandem colonoscopy. It consists of two withdrawal from the cecum to sigmoid colon using firstly High Definition White Light Endoscopy (WLE) and secondly Narrow Band Imaging (NBI). All detected polyps will be classified macroscopically and resected in each withdrawal.
  Interventions: Device: NBI; Device: WLE
- NBI-WLE (Experimental): Participants will be evaluated by same endoscopist, back-to-back tandem colonoscopy. It consists of two withdrawal from the cecum to sigmoid colon using firstly Narrow Band Imaging (NBI) and secondly High Definition White Light Endoscopy (WLE). All detected polyps will be classified macroscopically and resected in each withdrawal.
  Interventions: Device: NBI; Device: WLE

INTERVENTIONS:
Device: NBI — Withdrawal from cecum to sigmoid colon with Narrow Band Imaging (NBI, Evis Exera III, Olympus)
  Other Names: Narrow Band Imaging
Device: WLE — Withdrawal from cecum to sigmoid colon with High Definition White Light Endoscopy (WLE)
  Other Names: High Definition White Light Endoscopy

SUMMARY:
This study is designed to evaluate the utility of Narrow Band Imaging (NBI) compared with High Definition White Light colonoscopy (WLE) in subjects with serrated lesions who do not fulfill the diagnostic criteria of Serrated Polyposis Syndrome (SPS).

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of cancer death in western countries. Conventional polyps were considered the precursor lesions of all cases of sporadic colon cancer. Recently, serrated lesions and especially the Sessile Serrated Adenoma (SSA), are responsible of interval CRC between 20% to 35% of all CRC cases. These polyps are difficult to identify at endoscopy because they are located in the right colon, they are sessile or flat morphology and are pale color with mucus capping.

According to the WHO, SPS is defined with one of the following criteria: (1) at least 5 serrated polyps proximal to the sigmoid colon, 2 of which are greater than 10 mm in diameter; (2) any number of serrated polyps occurring proximal to the sigmoid colon in an individual who has a first-degree relative with serrated polyposis; or (3) more than 20 serrated polyps of any size distributed throughout the colon. Therefore, patients with SPS are considered to be at increased risk of CRC. Considering the substantial risk of polyp recurrence, it is mandatory to follow up an annual surveillance.

Narrow-Band Imaging (NBI, Olympus) selectively uses certain wavelengths of the visible light leading to a shift in the excitation spectrum towards blue light. Blood vessels will appear dark, allowing an improved visibility and identification of the surface and vascular structures. In contrast to conventional chromoendoscopy, it is easily activated by pressing a button on the endoscope. A pilot study in patients with SPS showed significantly lower polyp miss rate with NBI compared with WLE. Furthermore, the European Society of Gastrointestinal Endoscopy (ESGE) has recently published the first Guideline of Advanced Endoscopic Imaging for the detection and differentiation of colorectal neoplasia and recommends conventional chromoendoscopy or NBI in patients with SPS (strong recommendation, low quality evidence).

The hypothesis is that NBI could improve the detection rate of serrated polyps compared with WLE in patients who do not accomplish the SPS criteria.

The investigators will perform a randomised, cross-over trial of tandem colonoscopy using NBI and WLE. The main goal is to compare the rate of detected polyps between both techniques and, if it is necessary, reassessing the diagnosis for an appropriate surveillance interval.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 50 years old who accept CRC screening colonoscopy
* Patients with a basal colonoscopy findings: ≥1 serrated polyps proximal to the sigmoid colon, which are greater than ≥10mm in diameter; or ≥3 serrated polyps proximal to the sigmoid colon

Exclusion Criteria:

* Diagnosis of a CRC in the basal colonoscopy
* Subjects with other types of histology polyps
* Subjects who neglect to follow-up
* Subjects who do not accept informed consent
* Subjects with high risk of perforation or complications due to sedation, including patients with comorbidities (ASA IV-V)
* Inadequate bowel preparation for colonoscopy (defined by Boston Bowel Preparation Score (BBPS): ≤ 5 total points; or 0-1 points in any of the 3 segments of the colon)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of polyps detected with both techniques (NBI versus WLE) | Less than 1 year after the basal colonoscopy
  Efficacy of NBI in detecting serrated polyps compared with WLE

SECONDARY OUTCOMES:
Number of new patients who accomplish the SPS criteria | Less than 1 year after the basal colonoscopy
Number of missed lesions on basal colonoscopy | Less than 1 year after the basal colonoscopy
  Compare the number of missed lesions on the index examination based on the colonoscopy findings (NBI and WLE)
Number of accurate detection of adenomas with morphologic features with both groups (NBI and WLE) compared to histopathology | Less than 1 year after the basal colonoscopy
  Accuracy in detecting adenomas endoscopically compared with histopathology (gold standard)

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Riu, MD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Hospital del Mar, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ferlay J, Steliarova-Foucher E, Lortet-Tieulent J, Rosso S, Coebergh JW, Comber H, Forman D, Bray F. Cancer incidence and mortality patterns in Europe: estimates for 40 countries in 2012. Eur J Cancer. 2013 Apr;49(6):1374-403. doi: 10.1016/j.ejca.2012.12.027. Epub 2013 Feb 26. PMID 23485231
- [Result] Siegel R, Desantis C, Jemal A. Colorectal cancer statistics, 2014. CA Cancer J Clin. 2014 Mar-Apr;64(2):104-17. doi: 10.3322/caac.21220. Epub 2014 Mar 17. PMID 24639052
- [Result] Winawer SJ, Zauber AG, Ho MN, O'Brien MJ, Gottlieb LS, Sternberg SS, Waye JD, Schapiro M, Bond JH, Panish JF, et al. Prevention of colorectal cancer by colonoscopic polypectomy. The National Polyp Study Workgroup. N Engl J Med. 1993 Dec 30;329(27):1977-81. doi: 10.1056/NEJM199312303292701. PMID 8247072
- [Result] van Rijn JC, Reitsma JB, Stoker J, Bossuyt PM, van Deventer SJ, Dekker E. Polyp miss rate determined by tandem colonoscopy: a systematic review. Am J Gastroenterol. 2006 Feb;101(2):343-50. doi: 10.1111/j.1572-0241.2006.00390.x. PMID 16454841
- [Result] Brown SR, Baraza W. Chromoscopy versus conventional endoscopy for the detection of polyps in the colon and rectum. Cochrane Database Syst Rev. 2010 Oct 6;(10):CD006439. doi: 10.1002/14651858.CD006439.pub3. PMID 20927746
- [Result] Kaminski MF, Hassan C, Bisschops R, Pohl J, Pellise M, Dekker E, Ignjatovic-Wilson A, Hoffman A, Longcroft-Wheaton G, Heresbach D, Dumonceau JM, East JE. Advanced imaging for detection and differentiation of colorectal neoplasia: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2014 May;46(5):435-49. doi: 10.1055/s-0034-1365348. Epub 2014 Mar 17. PMID 24639382
- [Result] Boparai KS, van den Broek FJ, van Eeden S, Fockens P, Dekker E. Increased polyp detection using narrow band imaging compared with high resolution endoscopy in patients with hyperplastic polyposis syndrome. Endoscopy. 2011 Aug;43(8):676-82. doi: 10.1055/s-0030-1256447. Epub 2011 Aug 2. PMID 21811939
- [Result] Leggett B, Whitehall V. Role of the serrated pathway in colorectal cancer pathogenesis. Gastroenterology. 2010 Jun;138(6):2088-100. doi: 10.1053/j.gastro.2009.12.066. PMID 20420948
- [Derived] Riu Pons F, Andreu M, Naranjo D, Alvarez-Gonzalez MA, Seoane A, Dedeu JM, Barranco L, Bessa X. Narrow-band imaging and high-definition white-light endoscopy in patients with serrated lesions not fulfilling criteria for serrated polyposis syndrome: a randomized controlled trial with tandem colonoscopy. BMC Gastroenterol. 2020 Apr 16;20(1):111. doi: 10.1186/s12876-020-01257-4. PMID 32299380